CLINICAL TRIAL: NCT04714242
Title: Choroid and Choriocapillary Changes in Polypoidal Choroidal Vasculopathy After Intravitreal Anti-VEGF Therapy
Brief Title: OCTA and Polypoidal Choroidal Vasculopathy
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 1401/21
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Polypoidal Choroidal Vasculopathy
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients underwent anti-VEGF therapy: intravitreal Anti-VEGF therapy: Three monthly intravitreal injections
  Interventions: Drug: Ranibizumab Injection
- Control Group: Healthy eyes without actual and previous ocular diseases

INTERVENTIONS:
Drug: Ranibizumab Injection — Three monthly intravitreal injections of Ranibizumab
  Other Names: Lucentis
  Groups: Patients underwent anti-VEGF therapy

SUMMARY:
To investigate the structural and vascular features of choroid in patients affected by PCV after Ranibizumab intravitreal injection.

DETAILED DESCRIPTION:
Polypoidal choroidal vasculopathy represents a distinct form of choroidal neovascularization.

The study investigated the changes in choroidal vascular network after anti-VEGF therapy using optical coherence tomography angiography, a novel and non invasive diagnostic technique that allows to better understand the pathophysiologic mechanism of this neovascularization.

ELIGIBILITY:
Inclusion Criteria:

* age older than 60 years
* diagnosis of polypoidal choroidal vasculopathy
* absence of previous ocular surgery, congenital eye disease, high myopia (>6 dioptres), actual or previous diagnosis of glaucoma, optic disc anomaly, macular or vitreoretinal diseases.
* absence of significant lens opacities, low-quality OCT-A images.

Exclusion Criteria:

* age older than 80 years
* absence of diagnosis of polypoidal choroidal vasculopathy
* presence of previous ocular surgery, congenital eye disease, high myopia (>6 dioptres), actual or previous diagnosis of glaucoma, optic disc anomaly, macular or vitreoretinal diseases.
* presence of significant lens opacities, low-quality OCT-A images.

Ages: 60 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participans were older than 60 years with diagnosis of polypoidal choroidal vasculopathy They did not present other ophthalmological diseases.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Study of vascular features of choroid in polypoidal choroidal vasculopathy after intravitreal injections of Ranibizumab | 12 Months
  The effectiveness of Ranibizumab injections for treating PCV using optical optical coherence tomography angiography. The parameters analyzed by optical coherence tomography angiography were: choriocapillaris vessel density.

SECONDARY OUTCOMES:
Study of structural features of choroid in polypoidal choroidal vasculopathy after intravitreal | 12 Months
  The effectiveness of Ranibizumab injections for treating PCV using optical optical coherence tomography. The parameters analyzed by optical coherence tomography were: subfoveal choroidal thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy